CLINICAL TRIAL: NCT05870657
Title: Adherence and Persistence to Inclisiran Among Early Users in Germany
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839A12013
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: High Levels of Low-density Lipoprotein Cholesterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Overall cohort: Patients receiving inclisiran

SUMMARY:
The present study was a descriptive, non-interventional, retrospective cohort study aimed at evaluating early data on adherence, persistence, and treatment patterns among patients receiving inclisiran and other lipid-lowering therapies (LLT) in a real-world setting in Germany. Analysis was carried out using the IQVIA™ LRx database.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects ≥18 years old who were prescribed an inclisiran dose.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 1109 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with at least 5 months of potential follow-up who were prescribed a second dose of inclisiran | 8 months
Percentage of patients who were prescribed a second dose of inclisiran between 1 and 6 months after prescription of first dose | 8 months
Median time between first and second prescribed doses | 8 months

SECONDARY OUTCOMES:
Age and gender characteristics | 6 months
Age and gender distribution | 6 months
Prescriber specialty distribution for patients | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Basel, Switzerland